CLINICAL TRIAL: NCT00437619
Title: An Open Label Study to Evaluate the Clinical Response to Sequential Treatment With Daivobet and Daivonex in Patients With Mild to Moderate Psoriasis
Brief Title: A Study of Sequential Treatment With Daivobet (Betamethasone Dipropionate Plus Calcipotriol) and Daivonex (Calcipotriol) in Patients With Psoriasis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19876
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — calcipotriene

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: calcipotriol hydrate [Daivonex]

INTERVENTIONS:
Drug: calcipotriol hydrate [Daivonex] — 50 micrograms/g bid for 4 weeks (weeks 5-8) in patients who have shown a >50% response to Daivobet from weeks 0-4.

SUMMARY:
This single arm study will evaluate the efficacy and safety of sequential treatment with Diavobet (betamethasone propionate 0.5mg/g plus calcipotriol hydrate 50 micrograms/g) once daily for 4 weeks followed by Daivonex (calcipotriol hydrate 50 micrograms/g) twice daily for 4 weeks, in the control of signs and symptoms in patients with mild to moderate psoriasis. Only patients showing a >50% response to Daivobet will progress to the Daivonex maintenance phase. The anticipated time on study treatment is <3 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* clinical diagnosis of psoriasis vulgaris;
* PASI score 1-12 in >=1 body area.

Exclusion Criteria:

* clinical presentation of erythrodermic pustular psoriasis, expressed in plates and localized lesions on face and/or scalp;
* viral, fungal or bacterial skin infections;
* use of any topical treatment for psoriasis within previous 15 days;
* use of any systemic therapy and phototherapy for psoriasis within previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
PASI reduction | Weeks 4 and 8

SECONDARY OUTCOMES:
AEs. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Brazil (9):
  - Belém
  - Belo Horizonte
  - Botucatu
  - Brasília
  - Campinas
  - Curitiba
  - Rio de Janeiro
  - Salvador
  - São Paulo